CLINICAL TRIAL: NCT06120738
Title: The Effect Of Smartphone Addiction On Trunk Muscles Performance In Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ebrahim Elkomy, assistant lecturer, Cairo University
Other Study IDs: P.T.REC/012/004453
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-03

CONDITIONS: Smartphone Addiction; Muscle Weakness Condition; Adolescents
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- smartphone addiction group: smartphone addiction will be assessed using smartphone addiction scale short version(SAS-SV) evaluation of trunk muscles performance using isokinetic dynamometer

SUMMARY:
Statement of the problem:

Does overuse of the smartphones affect trunk muscles performance in normal adolescents it will be assumed that There will be no affection of smartphone addiction on trunk muscles performance in normal adolescents

DETAILED DESCRIPTION:
* Subjects:

  - Sixty - six normal healthy adolescent from both genders will be recruited for the study from high school students and first year university students, they will be divided according to their smart phone addiction scale short version (SAS-SV) scores into two groups: Group (A): smartphone addicts (consists of 33 participants) Group (B): smartphone non- addicts (consists of 33 participants)
* Inclusion criteria

  * Age ranges from 14 to 18 years
  * Have Body Mass Index (BMI) = 5th percentile to less than the 85th percentile 2. Exclusion criteria

Subjects will be excluded from the study if he/she has:

* visual or hearing defects
* overweight or obese
* neurological disorder
* marked musculoskeletal problem

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 14 to 18 years
* Have Body Mass Index (BMI) = 5th percentile to less than the 85th percentile

Exclusion Criteria:

* Subjects will be excluded from the study if he/she has:
* visual or hearing defects
* overweight or obese
* neurological disorder
* marked musculoskeletal problem

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Sixty - six normal healthy adolescent from both genders will be recruited for the study from high school students and first year university students, they will be divided according to their smart phone addiction scale short version (SAS-SV) scores into two groups:
  Group (A): smartphone addicts (consists of 33 participants) Group (B): smartphone non- addicts (consists of 33 participants)
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
evaluation of the trunk muscles performance | baseline only
  the isokinetic dynamometer will be used to assess the trunk muscles performance by using HUMAC CSMI isokinetic dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Aya Elkomy, PHD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - the Governement'S Secondary School and Universities, Tanta
  - the Governement'S Secondary Schools and Universities, Tanta

IPD SHARING:
Plan to Share IPD: Undecided